CLINICAL TRIAL: NCT00776269
Title: Comparison the Result of Argon Laser and Radiofrequency in Trichiasis Treatment of Patients Referred to Labbafinejad Oculoplastic Clinic
Brief Title: Comparison of Argon Laser and Radiofrequency in Trichiasis Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Ophtalmic Research Centre (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8724
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-09

CONDITIONS: Trichiasis
Keywords: Argon laser; Trichiasis; Radiofrequency; Patients with trichiasis
MeSH Terms: conditions — Trichiasis | interventions — Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- argon laser (Experimental)
  Interventions: Procedure: argon laser and radiofrequency

INTERVENTIONS:
Procedure: argon laser and radiofrequency

SUMMARY:
In this clinical trial study,the investigators intend to compare two methods of trichiasis treatment.One by argon laser and the other by radiofrequency then compare the result of these procedures, especially, the investigators would like to compare which of these have less complications such as bleeding,pain,notch in the site of surgery and etc.

ELIGIBILITY:
Inclusion Criteria:

* All patients who came to labbafinejad oculoplastic clinic due to trichiasis

Exclusion Criteria:

* Having a history of entropion
* Any history of previous laser ,radiofrequency therapy or surgery
* More than 50% of the area is involved with trichiasis
* More than 10 eye lashes need to be treated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2008-10

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran